CLINICAL TRIAL: NCT01141868
Title: Evaluating an Internet-based Intervention for Insomnia in Breast Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never opened due to technical upgrades that were needed for the SHUTi computer system.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Jane Schubart, PhD, Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 31944EP
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2010-06

CONDITIONS: Insomnia; Breast Cancer
Keywords: insomnia; breast cancer survivor; Internet intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Breast Neoplasms | interventions — Patient Portals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet Intervention (Experimental)
  Interventions: Behavioral: Internet Intervention
- Delayed Intervention (Experimental): Receive access to the online Internet intervention after completing post-assessments.
  Interventions: Behavioral: Internet Intervention

INTERVENTIONS:
Behavioral: Internet Intervention — online treatment for insomnia
  Other Names: Internet

SUMMARY:
This study examines the efficacy of an Internet-delivered intervention to reduce symptoms of insomnia in breast cancer survivors. Breast cancer patients with insomnia (N=30) will be assigned to either gain access to the 6-week treatment program immediately (experimental group) or following study participation (control group).

ELIGIBILITY:
Inclusion criteria:

* Female
* Diagnosed with breast cancer
* Age 18 and older
* Completed primary treatment at least one month prior to enrollment
* Diagnosis of insomnia

Exclusion criteria:

* Experiencing a sleep disorder other than insomnia (e.g., sleep apnea)
* Experiencing a major depressive episode or other serious psychiatric disturbance
* Modification of psychotropic medications within the previous month
* Undergoing current psychotherapy treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
sleep efficiency | 6 weeks
  sleep-onset latency, wake after sleep onset, and number of awakenings

SECONDARY OUTCOMES:
total sleep time | 6 wks
  total hours of sleep per 24 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Jane Schubart, PhD, Principal Investigator — Penn State